CLINICAL TRIAL: NCT05268354
Title: Modification of Characteristics Associated With the Noncontact Knee Injury Mechanism in Adult Recreational Netball Players
Brief Title: Modification of Risk Factors Associated With Knee Injury in Netball
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: St Mary's University College (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: StMarysUC2
Record Dates: First submitted 2022-02-24; First posted 2022-03-07 (Actual); Last update posted 2022-03-07 (Actual); Status verified 2022-02

CONDITIONS: Knee Injuries
MeSH Terms: conditions — Knee Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Training group (Experimental): 6-week neuromuscular training program
  Interventions: Other: 6-week neuromuscular training program
- Control group (No Intervention)

INTERVENTIONS:
Other: 6-week neuromuscular training program — Training program consisting of three neuromuscular training sessions per week
  Arms: Training group

SUMMARY:
Noncontact knee injuries are a concern in netball. As such, it is important to devise appropriate injury prevention programs that players will complete to reduce the risk of injury. Previous research suggests that the most common situation of noncontact knee injury in netball involves a stiff landing or apparent knee valgus collapse, trunk rotation, and lateral flexion. Therefore, the aim of this study is to investigate the effect of a neuromuscular training program on biomechanical risk factors during a netball-specific landing.

ELIGIBILITY:
Inclusion Criteria:

* Female
* 18-45 years
* No history of lower limb injury in the last 6 months
* No history of concussion in the last 6 months
* No history of any knee surgery
* Currently playing recreational netball at least once per week

Exclusion Criteria:

* Male
* Under 18 years or over 45 years of age
* Suffered from a lower limb injury in the last 6 months
* Suffered from concussion in the last 6 months
* Any history of knee surgery
* Not currently playing recreational netball at least once per week

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-03-04 (Estimated); Primary Completion 2024-01-31 (Estimated); Study Completion 2024-01-31 (Estimated)

PRIMARY OUTCOMES:
Peak knee flexion angle | From baseline to end of six-week training program
  Maximum angle of knee flexion on landing from a jump
Peak vertical ground reaction force | From baseline to end of six-week training program
  Maximum vertical ground reaction force on landing from a jump
Joint position sense | From baseline to end of six-week training program
  Ability to recreate knee angle in a seated position
Peak hamstring torque | From baseline to end of six-week training program
  Maximum isometric hamstring torque
Peak quadriceps torque | From baseline to end of six-week training program
  Maximum isometric quadriceps torque
Peak hip abductor torque | From baseline to end of six-week training program
  Maximum isometric hip abductor torque
Time to stabilization | From baseline to end of six-week training program
  Time to stabilization following landing from a jump
Peak horizontal jump distance | From baseline to end of six-week training program
  Maximum distance covered in a horizontal jump

IPD SHARING:
Plan to Share IPD: No